CLINICAL TRIAL: NCT05165563
Title: Comparison of Treatment Time Between Digital and Conventional Workflows for Treatment With Posterior Implant Restorations
Brief Title: Treatment Time Comparing Digital & Conventional Workflows
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Align Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-DT/PY-IRB 2020/DT010
Record Dates: First submitted 2021-11-22; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Dental Implant
Keywords: Clinical Research; Dental Implant; Digital Workflow; Crowns; Treatment time

STUDY DESIGN:
Intervention Model Description: Digital and conventional workflows for treatment of implant single crowns, and also the material used.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workflows (Experimental): Digital and conventional workflows for treatment of implant single crowns
  Interventions: Procedure: Treatment of implant single crown
- Materials (Experimental): Materials for treatment of implant single crowns (polymer-infiltrated ceramic networks, PICNs and lithium disilicate, LS2).
  Interventions: Procedure: Treatment of implant single crown

INTERVENTIONS:
Procedure: Treatment of implant single crown — Digital or Conventional Workflows for treatment of implant single crown and materials used.

SUMMARY:
This randomized controlled trial (RCT) analyzed monolithic single-unit implant restorations out of lithium disilicate (LS2) or polymer-infiltrated ceramic networks (PICN) in a chairside digital workflow (Test) and a conventional protocol (Control). The primary outcome was to investigate the treatment time of the overall operation. The null hypothesis of this RCT was that both workflows had comparable results with respect to the defined outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The participants having a transmucosal implant system (Straumann TL RN/WN, Institut Straumann, AG, Basel, Switzerland) were placed in a single-tooth gap in the area of premolar or molar regions in the maxilla and mandible with existing interproximal and antagonist contacts.
* general medical health is healthy or has a well-controlled systemic disease.
* general oral health has shown no sign of infection or unsuccessfully treated diseases such as chronic periodontitis.

Exclusion Criteria:

* smoking more than 10 cigarettes per day.
* pregnancy.
* psychiatric disorder
* history of radiation therapy at the head and neck area.
* history of chemotherapy.
* history of bony pathologies such as osseous dysplasia, odontogenic cyst or tumor, etc.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Treatment time | First visit to prosthesis delivery visit, through study completion, an average of 1 month
  Treatment time in every steps were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joda T, Bragger U. Time-Efficiency Analysis Comparing Digital and Conventional Workflows for Implant Crowns: A Prospective Clinical Crossover Trial. Int J Oral Maxillofac Implants. 2015 Sep-Oct;30(5):1047-53. doi: 10.11607/jomi.3963. PMID 26394340